CLINICAL TRIAL: NCT01149460
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Valacyclovir 1000 mg Tablet and Valtrex Administered as 1 x 1000 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Valacyclovir 1000 mg Tablet Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 40280
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Experimental): Test 1000 mg Tablet
  Interventions: Drug: Valacyclovir
- Valtrex (Active Comparator): Reference Listed Valacyclovir 1000 mg Tablet
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — Test 1000 mg Tablet
  Arms: Valacyclovir
Drug: Valacyclovir — Reference Listed Valacyclovir 1000 mg Tablet
  Other Names: Valtrex
  Arms: Valtrex

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Teva Pharmaceuticals USA valacyclovir and GlaxoSmithKline, USA (Valtrex) valacyclovir, administered as 1 x 1000 mg tablet under fed conditions.

ELIGIBILITY:
Inclusion Criteria

* Male or female, non-smokers, 18 years of age and older.
* Capable of consent

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses or surgery within 4 weeks of the administration of study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* BMI less than 19.0 or greater than or equal to 30.0 kg/m2.
* History of significant alcohol abuse within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40% alcohol]) or positive urine drug screen at screening.
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, valacyclovir, acyclovir, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to the administration of the study medication.
* Use of an investigational drug or participation in an investigation study within 30 days prior to the administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 90 days preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, could contraindicate the subjects participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Intolerance to venipunctures.
* Clinically significant history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Unable to understand or unwilling to sign the Informed Consent Form.
* Breast-feeding.
* Positive urine pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception:
* Intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration),
* Condom or diaphragm + spermicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Valacyclovir: Test 1000 mg Tablet dosed in first period follwed by Reference Listed 1000 mg Valtrex® tablet in second period
- Valtrex®: Reference Listed Valtrex® 1000 mg Tablet dosed in first period followed by Test 1000 mg Valacyclovir tablet in second period
Period: Overall Study
Arm/Group | Valacyclovir | Valtrex®
Started | 18 | 18
Completed | 18 | 16
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Valtrex® | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma) - Valacyclovir
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 12 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng/mL | 385.35 (139.10) | 350.86 (133.20)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of Least Squares Means (T/R) = 111.34, 90% CI 2-sided [100.54 to 123.29] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the test (T) and reference (R) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration) - Valacyclovir
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 12 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng*h/mL | 549.32 (137.87) | 551.77 (140.73)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means (T/R) = 100.01, 90% CI 2-sided [96.34 to 103.82] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity) - Valacyclovir
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 12 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng*h/mL | 552.17 (138.76) | 554.53 (140.97)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means (T/R) = 100.01, 90% CI 2-sided [96.38 to 103.78] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma) - Acyclovir
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng/mL | 6485.51 (1469.43) | 6283.25 (1375.42)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means (T/R) = 103.48, 90% CI 2-sided [97.87 to 109.41] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: AUC0-t (Area Under Concentration-time Curve From Time Zero to Time of Last Measurable Concentration) - Acyclovir
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng*h/mL | 22514.36 (4316.76) | 22675.85 (4063.20)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means (T/R) = 99.20, 90% CI 2-sided [97.14 to 101.31] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity) - Acyclovir
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Valacyclovir | Valtrex®
Number analyzed (Participants) | 18 | 16
ng*h/mL | 22705.17 (4336.16) | 22887.99 (4065.19)
Statistical Analysis 1: Comparison: Valacyclovir vs Valtrex®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 99.10, 90% CI 2-sided [97.04 to 101.19] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Valacyclovir | Valtrex®
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 7/36 | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=36) | Valtrex® (N=36)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Abdominal Pain/Cramp (Gastrointestinal disorders) | 0 (0) | 4 (4)
Loose/Soft Stools (Gastrointestinal disorders) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Low Hemoglobin Level (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Fatigue/Drowsiness (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.